CLINICAL TRIAL: NCT04406467
Title: Retrospective Review of Xen Gel Stent Implantation With Open vs. Closed Conjunctiva Approach
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00201210; 133133 (Other Grant/Funding Number: Allergan Inc.)
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2020-08

CONDITIONS: Glaucoma, Open-Angle
Keywords: Glaucoma surgery; Xen Gel Stent
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Xen Gel Stent — Ab-interno or Ab-Externa Xen with closed or open conjunctiva.

SUMMARY:
To measure surgical success of open vs closed conjunctiva with Xen implantation.

DETAILED DESCRIPTION:
This retrospective, single-arm multicenter study included >100 eyes (>100 patients) with glaucoma refractory to medical therapy. All surgeries were performed by two groups of surgeons at Johns Hopkins University and the sub-investigator group at New York University. Group 1: Xen with open conjunctiva for positioning and application of mitomycin. The Xen was placed through the sclera either ab-interno or ab-externa. Group 2 had Xen placed ab-interno or ab-externa (trans conjunctival), but the conjunctiva was not opened for positioning or application of mitomycin-C.

Success rates will be determined based on need for re-intervention and intraocular pressure control.

ELIGIBILITY:
Inclusion Criteria:

* Require surgery for uncontrolled glaucoma

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to the two institutions with elevated IOP and required surgery to lower IOP.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2017-11-19 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
re-intervention rate | 3 months
  This will be assessed as the proportion of patients that will need fibrosis relief by stent re-implantation

SECONDARY OUTCOMES:
Change in intraocular pressure | 1 day, 1 week, 1 month and 3 months
  will be assessed as a % change in intraocular pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Univeristy, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
De-identified internal use data.

REFERENCES:
- [Background] Panarelli JF, Yan DB, Francis B, Craven ER. XEN Gel Stent Open Conjunctiva Technique: A Practical Approach Paper. Adv Ther. 2020 May;37(5):2538-2549. doi: 10.1007/s12325-020-01278-1. Epub 2020 Mar 21. PMID 32200534
- [Derived] Do A, McGlumphy E, Shukla A, Dangda S, Schuman JS, Boland MV, Yohannan J, Panarelli JF, Craven ER. Comparison of Clinical Outcomes with Open Versus Closed Conjunctiva Implantation of the XEN45 Gel Stent. Ophthalmol Glaucoma. 2021 Jul-Aug;4(4):343-349. doi: 10.1016/j.ogla.2020.12.003. Epub 2020 Dec 13. PMID 33321200